CLINICAL TRIAL: NCT05107661
Title: Colorectal Screening Strategies in the High Risk Medically Underserved Population in a Hospital-based Community Outreach Program
Brief Title: Colorectal Screening Strategies in Underserved Populations
Status: Terminated | Type: Observational
Why Stopped: Preliminary findings revealed to many barriers to successfully complete this trial.
Sponsor: Virtua Health, Inc. (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-2021-03
Record Dates: First submitted 2021-10-05; First posted 2021-11-04 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Telephone Prompt: Following consent, the Research Team will call participants three times in the first month (within the first week of signing consent at week 2 and repeated at week 3) and then one time per month for the following two months with scripted messaging reminding the participant to complete the screening activity (colonoscopy or fecal test). Interpreter services via phone will be utilized for non-English speaking participants.
  Interventions: Behavioral: Telephone Prompt
- Digital Prompt: Following consent, scripted messaging will be sent three times in the first month (within the first week of signing consent at week 2 and repeated at week 3) and then once time per month for the following two months with scripted messaging reminding the participant to complete the screening activity (colonoscopy or fecal test). Digital prompts will be available in Spanish and English.
  Interventions: Behavioral: Telephone Prompt

INTERVENTIONS:
Behavioral: Telephone Prompt — Scripted messaging to remind subjects to complete their colorectal screening (colonoscopy or fecal test)
  Other Names: Digital Prompt

SUMMARY:
Research efforts are necessary to identify strategies to increase colorectal screening in underserved patient populations. Racial, ethnic minorities and medically underserved individuals continue to experience disparities in colorectal cancer mortality despite the availability of screening tests that can detect tumors early when treatments are most effective.

DETAILED DESCRIPTION:
To determine the effectiveness of completion of colorectal cancer screening through fecal testing for blood and/or colonoscopies as a screening intervention utilizing digital reminders versus telephone prompts and reminders in economically disadvantaged minority communities as part of a colorectal screening outreach program.

ELIGIBILITY:
Inclusion Criteria:

* Any Gender
* 45-64 years of age
* Able to sign the informed consent form
* Meets eligibility criteria to participate in New Jersey Cancer Education Early Detection Community Outreach Program

  * Uninsured/underinsured
  * Household income <250% Federal Poverty Level
  * Must be New Jersy resident
* Must have Smart phone
* Must speak English or Spanish

Exclusion Criteria:

* History of colon cancer, colon/rectal polyps and rectal bleeding
* Individuals with Dementia
* ECOG Performance Status 3-4
* Prior Colonoscopy within past 10 years

Ages: 45 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: The target population is economically disadvantaged minority, medically underserved individuals that meet eligibility requirements for participation in the New Jersey Cancer Education Early Detection Program.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
: Colorectal Screening Strategies in the High Risk Medically Underserved Population in a Hospital-based Community Outreach Program | 3 month intervals
  To determine the effectiveness of digital reminders versus telephone reminders to prompt participants to follow through with completing their colonoscopy. Comparison of the success or failure of digital versus phone call reminders will be measured. To determine the effectiveness of digital reminders versus phone reminders to follow through with completing fecal testing to screen for colorectal cancer. Comparison of the success or failure of digital versus phone call reminders will be measured.

SECONDARY OUTCOMES:
Colorectal Screening Strategies in the High Risk Medically Underserved Population in a Hospital-based Community Outreach Program | 3 month intervals
  Which colorectal screening intervention is preferred in the target population: Colonoscopy versus occult fecal testing in the targeted population
  * Out comes will be measured by:
  * Percentage rates of which screening method is selected by the participant: colonoscopy vs. fecal testing.
  * Percentage rates for following through with completing the screening colonoscopy versus occult fecal testing in the targeted population

CONTACTS AND LOCATIONS:
Locations (1):
- Virtua Health, Voorhees Township, New Jersey, United States